CLINICAL TRIAL: NCT06535932
Title: An Assessment of Patient Preference for the Amara View Full Face Mask Compared to the ResMed AirFit F40 -a Benchmark Protocol
Brief Title: Amara View Benchmark Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SRC-300401-Amara ViewBenchmark
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Results first posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Sleep Apnea Syndromes
Keywords: Positive Airway Pressure Therapy; Minimal contact full face mask
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: Randomized crossover
Masking Description: N/A - No masking will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Amara View Minimal Contact Full Face Mask (Active Comparator): Participants will wear the Amara View mask for 15 days
  Interventions: Device: Amara View Minimal Contact Full Face Mask
- F40 Minimal Contact Full Face Mask (Active Comparator): Participants will wear the F40 for 15 days
  Interventions: Device: F40 Minimal Contact Full Face Mask

INTERVENTIONS:
Device: Amara View Minimal Contact Full Face Mask — The Amara View Full-Face Mask is a minimal contact full face mask manufactured by Philips Respironics (Murrysville, PA) that covers the mouth and seals under the nose compared to traditional full-face masks which seal over the nose. The Amara View mask is intended to reduce discomfort on the bridge of the nose. There is no forehead arm, offering patients an enhanced design to keep the field of vision clear.
  Arms: Amara View Minimal Contact Full Face Mask
Device: F40 Minimal Contact Full Face Mask — The AirFit F40 is a minimal contact FFM manufactured by ResMed (San Diego, CA) that rests softly and securely under the patients nose and is designed to let patients sleep in any position and move freely throughout the night. The mask consists of three cushion sizes and three headgear sizes. Headgear adjustments can be made with magnetic clips that easily snap on and off.
  Arms: F40 Minimal Contact Full Face Mask

SUMMARY:
This randomized crossover, benchmark clinical trial aims to compare the Philips Amara View and ResMed AirFit F40 minimal contact full face masks on patient preference of mask attributes and usage parameters. At the first study visit participants will be fitted with either the Amara View or the AirFit F40. The order in which participants will use the masks will be randomized. After the fitting and completion of informed consent, eligibility, and baseline questionnaires, participants will take home the first mask and use it with their prescribed PAP device for 15-days. After the first 15-day time period participants will return for their second visit. At this visit participants will return the first mask to the study team and complete a survey on the mask attributes. They will then be fitted with the second study mask and will be given the mask to take home and use with their prescribed PAP device for 15-days. At the end of the second 15-day trial period, participants will return for the third study visit. At this visit they will return the second mask and complete a mask attributes survey on the second mask.

DETAILED DESCRIPTION:
Participants will be recruited via a sleep clinic contracted to recruit participants within the United States. Study staff will be responsible for assessment of inclusion and exclusion criteria. Scheduling will be conducted by the site. Participants who are willing to enroll will be scheduled for an in-person visit to provide informed consent and complete study procedures. During the baseline visit, review the Informed Consent Form (ICF) with the participant explaining and answering any questions the participant may have about the study. If the participant is willing to take part in the study, the ICF will be signed and dated by the participant and the site study representative obtaining consent. Those who provide consent will then complete the Demographics Questionnaire, Baseline Mask Survey, and Eligibility Questionnaire to confirm entry criteria. Participants will be asked to bring their prescribed mask and PAP device to Visit 1.At the initial visit, participants will undergo a fitting of the mask they are randomized to start the study with; either the Amara View or the AirFit F40 mask. Participants will be fit with mask sizes recommended by the clinician. The clinician will use the provided sizing gauges for the Amara View and AirFit F40 masks respectively. Once a mask size is selected for the first study mask, the participant will undergo short trials using his or her own PAP machine at therapeutic pressure, and an assessment of mask fit will be performed. If the participant's PAP device is not available, they will be fitted with the mask and will undergo short trials using a PAP device provided by the site. Participants may be fitted with up to three mask sizes for the mask. A Mask Fitting Survey will be used to capture the participant's prescribed pressure, mask (cushion/frame) sizes and fitting observations for the first study mask.

After the mask fitting, participants will be given the first study mask to take home. They will be encouraged to use the mask for the full 15-days of the first trial period. After the first 15-day trial period with the first study mask, participants will return to the site for their second study visit. Participants will be instructed to bring their PAP device and the first study mask to the visit. Participants will complete a mask attributes survey on the first study mask and then they will be fitted with the second study mask. Fitting procedures will follow the same procedure as described above in the baseline visit. After the mask fitting, participants will be given the second study mask to take home. They will be encouraged to use the mask for the full 15 days of the second trial period. After the second 15-day trial period with the second study mask, participants will return to the site for the third and final study visit. During this visit, participants will complete a mask-attributes survey on the second study mask and return all study product.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21-85 years (inclusive)
* Weight >66 pounds/30 kg
* Established on PAP for ≥90 days at the time of consent
* Currently prescribed and using fixed pressure, Auto CPAP, or Bi-Level therapy on a regular basis (average PAP usage of ≥4 hours/night, ≥ 4 days per week for ≥3 months)
* Currently using a Full-Face mask
* Able to read, write, speak and understand English
* Willing and able to provide informed consent
* Willing and able to follow instructions and complete all activities required by the study
* Able to remove a sleep apnea mask without assistance

Exclusion Criteria:

* Currently using a Philips Respironics Amara View FFM or ResMed AirFit F40 FFM
* Allergy to silicone
* Allergy to latex
* Unique facial features (i.e., deformities of the face and/or head, piercings, etc.) that could interfere with the therapeutic use of this type of mask
* Employee or living with a family member who works for Philips or any company that designs, sells, or manufactures sleep-related products.
* Prescribed oxygen at night or continuously
* Recent eye surgery or dry eyes
* Hiatal hernia
* Excessive reflux
* Impaired cough reflux
* Impaired cardiac sphincter function
* Using prescription drugs that induce vomiting
* Currently participating in another interventional research study or planned participation in another interventional clinical research study during the trial period
* Prescribed an ASV (adaptive servo-ventilation) device
* Prescribed mechanical ventilation
* Pre-existing conditions such as bullous lung disease, pathologically low blood pressure, bypassed upper airway, pneumothorax, pneumocephalus, cerebral spinal fluid (CSF) leaks, or cribriform plate abnormalities
* Any unstable medical condition (e.g., uncontrolled cardiac, lung, or neurological disease) or limitation that would affect the participant's ability to complete trial activities
* Experiencing any acute illness (e.g., acute sinusitis, ear or eye infections, upper respiratory infections, pharyngitis, bronchitis, pleurisy, pneumonia, or facial dermatitis) that would impact their ability to use the mask and/or PAP therapy during the trial
* Surgical procedures involving the head, neck, face (eyes, ears, nose), or lungs in the previous 90 days or taking place any time during the trial period
* Pregnant
* Advised by a health care provider to avoid magnets
* Patient or patient's household member, caregiver or bed partner in close vicinity currently using medical implants or medical devices that would be affected by magnets, including but not limited to:

  * Pacemakers
  * Implantable cardioverter defibrillators (ICD)
  * Neurostimulators
  * Magnetic metallic implants/electrodes/valves placed in upper limbs, torso, or higher (i.e., neck and head)
  * Cerebral spinal fluid (CSF) shunts (e.g., ventriculo peritoneal (VP) shunt)
  * Aneurysm clips
  * Embolic coils
  * Intracranial aneurysm intravascular flow disruption devices
  * Metallic cranial plates, screws, burr hole covers, and bone substitute devices
  * Metallic splinters in the eye
  * Ocular implants (e.g., glaucoma implants, retinal implants)
  * Certain contact lenses with metal
  * Implants to restore hearing or balance that have an implanted magnet (such as cochlear implants, implanted bone conduction hearing devices, and auditory brainstem implants)
  * Magnetic denture attachments
  * Metallic gastrointestinal clips
  * Metallic stents (e.g., aneurysm, coronary, tracheobronchial, biliary)
  * Implantable ports and pumps (e.g., insulin/infusion pumps)
  * Hypoglossal nerve stimulators
  * Devices labeled as MR (Magnetic Resonance) unsafe
  * Magnetic metallic implants not labeled for MR or not evaluated for safety in a magnetic field
* PAP device is unknown, or they are using a recalled device that has not yet been remediated. Recalled devices include:

  * DreamStation CPAP, Auto CPAP, or BiPAP
  * DreamStation BiPAP, autoSV (ASV)
  * DreamStation ST, AVAPS (Also known as DreamStation BiPAP AVAPS or DreamStation BiPAP S/T)
  * DreamStation Go CPAP, APAP or Auto CPAP
  * Dorma 400 or 500 CPAP or Auto CPAP
  * System One ASV4
  * System One (Q-Series) 50 series CPAP, Auto CPAP, or BiPAP
  * System One (Q-Series) 60 series CPAP, Auto CPAP, or BiPAP
  * C Series ASV, S/T, or AVAPS
  * REMStar SE Auto CPAP

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2024-07-25 (Actual); Primary Completion 2024-09-06 (Actual); Study Completion 2024-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Ojile, MD, Principal Investigator — Clayton Sleep Institute
Locations (1):
- Clayton Sleep Institute, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Amara View First, Then ResMed AirFit F40: Participants wore the Amara View mask for the first15 days, then wore the ResMed Airfit F40 for the second 15 days.
- ResMed AirFit F40 First, Then Philips Amara View: Participants wore the AirFit F40 for the first 15 days, then the Amara View for the second 15 days.
Period: Overall Study
Arm/Group | Amara View First, Then ResMed AirFit F40 | ResMed AirFit F40 First, Then Philips Amara View
Started | 16 | 19
Completed | 16 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants were enrolled and randomized.
Arm/Group | All Participants
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (9.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 20
  Female | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 33
  More than one race | 0
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino/a | 1
  Not Hispanic or Latino/a | 33
  Not Known or not reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Patient Preference on Mask Attributes
Description: Comparison in satisfaction ratings between the Amara View and the AirFit F40 on mask attributes including:
  bed partner satisfaction, fit, comfort, ability to maintain a seal during use, stability of the mask, noise level, air venting, comfort of breathing, sleep quality, visual appeal, and overall satisfaction. The scale for each mask attribute ranges from 0 to 10, where 0 indicates the lowest satisfaction and 10 indicates highest satisfaction. Each mask attribute was rated and analyzed individually; the scores from the separate mask attributes were not totaled.
Time Frame: up to 35 days
Population: All 35 participants tried both masks in randomized order.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Amara View Minimal Contact Full Face Mask | F40 Minimal Contact Full Face Mask
Number analyzed (Participants) | 35 | 35
scores on a scale
  Bed partner satisfaction | 5.6 (3.87) | 7.07 (3.35)
  Fit | 7.66 (2.63) | 7.66 (2.53)
  Comfort | 7.2 (2.85) | 7.34 (3.02)
  Ability to maintain a seal during use | 6.66 (3.14) | 7.03 (3.26)
  Stability of the mask | 7.03 (3.25) | 6.51 (3.45)
  Noise level | 7.34 (3.16) | 8.43 (2.34)
  Air venting | 7.71 (2.64) | 9 (1.68)
  Comfort of breathing | 8.49 (2.34) | 8.43 (2.48)
  Sleep quality | 6.86 (3.42) | 7.11 (3)
  Visual appeal | 8.89 (1.37) | 8.91 (1.36)
  Overall satisfaction | 6.17 (3.34) | 6.69 (2.85)

2. Primary Outcome: Ease of Use
Description: Ease of use and satisfaction ratings between the Amara View and the AirFit F40 on the following parameters: mask clips, mask overall, assembly, disassembly. The scale for each ease-of-use attribute ranges from 0 to 10, where 0 indicates the most difficult and 10 indicates the easiest. Each ease-of-use attribute was rated and analyzed individually; the scores from the separate attributes were not totaled.
Time Frame: up to 35 days
Population: All 35 participants tried both masks in randomized order.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Amara View Minimal Contact Full Face Mask | F40 Minimal Contact Full Face Mask
Number analyzed (Participants) | 35 | 35
scores on a scale
  Overall Ease of Use | 7.09 (2.57) | 8.46 (2.15)
  Mask clips | 7.73 (2.63) | 8.79 (1.63)
  Ease of attaching cushion | 9.1 (1.41) | 8.8 (2.44)
  Ease of removing cushion | 8.87 (1.51) | 9.2 (1.42)

3. Primary Outcome: Difference in Net Promotor Score
Description: Difference in the Net Promotor Score between the Amara View and AirFit F40. The Net Promotor score is based on a 0 to 10 scaled question "Would you recommend this (Amara View FFM or AirFit F40) mask to others?" where 0 indicates "unlikely to recommend" and 10 indicates "likely to recommend". The 0 to 10 scale is grouped into three categories: promoters (ratings 9-10), detractors (ratings 0-6), and neutral (7-8). Net Promoter Scores (NPS) were calculated by subtracting the percentage of detractors from the percentage of promoters: [% Promoters] - [% Detractors]. Ratings of 7-8 were considered neutral. The NPS scale ranges from -100 to 100. Scores less than 100 indicate that the percentage of detractors exceeds the percentage of promoters. Scores greater than 100 indicate the percentage of promoters exceeds the percentage of detractors. A NPS score of 0 indicates the percentages of promoters and detractors are equal.
Time Frame: Up to 35 days
Measure: Number (95% Confidence Interval); unit: scores on a scale
Arm/Group | Amara View Minimal Contact Full Face Mask | F40 Minimal Contact Full Face Mask
Number analyzed (Participants) | 35 | 35
scores on a scale | -28.6 [-54.3 to -2.8] | -11.4 [-38.6 to 15.7]

4. Primary Outcome: Patient Preference
Description: Percentage of patients who prefer the Amara View compared to the AirFit F40 for the following: seal, comfort, stability, noise level, headgear, mask cushion ease of use, less disruptive air venting, and overall preference.
Time Frame: Up to 35 days
Population: The below percentages may not total 100 because some participants indicated no preference.
Measure: Count of Participants; unit: Participants
Arm/Group | Amara View Minimal Contact Full Face Mask | F40 Minimal Contact Full Face Mask
Number analyzed (Participants) | 35 | 35
Participants
  Seal | 12 | 17
  Comfort | 10 | 19
  Stability | 12 | 14
  Noise level | 4 | 16
  Headgear | 8 | 17
  Mask cushion ease of use | 4 | 10
  Less disruptive air venting | 2 | 14
  Overall preference | 9 | 20

5. Secondary Outcome: Leak
Description: Comparison of leak values between the Amara View and F40.
Time Frame: up to 35 days
Population: Data only available from the four participants who used a Philips PAP device.
Measure: Mean (Standard Deviation); unit: liters per minute
Arm/Group | Amara View Minimal Contact Full Face Mask | F40 Minimal Contact Full Face Mask
Number analyzed (Participants) | 4 | 4
liters per minute | 37.4 (10.3) | 40.6 (15.3)

6. Secondary Outcome: Number of Sleep Apnea Events Per Hour Measured by the Residual Apnea Hypopnea Index (AHI)
Description: Comparison of residual Apnea Hypopnea Index (AHI) between the Amara View and F40. Residual AHI refers to the remaining or persistent apnea-hypopnea index (AHI) after a patient has undergone treatment, typically continuous positive airway pressure (CPAP) therapy, for obstructive sleep apnea (OSA). It represents the number of apnea and hypopnea events per hour of sleep that still occur despite treatment.
Time Frame: up to 35 days
Population: Data only available from the four participants who used a Philips PAP device.
Measure: Mean (Standard Deviation); unit: events per hour
Arm/Group | Amara View Minimal Contact Full Face Mask | F40 Minimal Contact Full Face Mask
Number analyzed (Participants) | 4 | 4
events per hour | 3.27 (1.1) | 3.85 (0.98)

7. Secondary Outcome: Air Pressure
Description: Air pressure (cmH20) used during PAP therapy while using the Amara View and AirFit F40 masks.
Time Frame: 30 days
Population: Data only available from the four participants who used a Philips PAP device.
Measure: Mean (Standard Deviation); unit: cmH20
Arm/Group | Amara View Minimal Contact Full Face Mask | F40 Minimal Contact Full Face Mask
Number analyzed (Participants) | 4 | 4
cmH20 | 10.6 (2.38) | 11.3 (2.71)

8. Secondary Outcome: Adherence to PAP Therapy
Description: Daily hours of use of PAP therapy while using the Amara View and AirFit F40 masks.
Time Frame: up to 35 days
Population: Data only available from the four participants who used a Philips PAP device.
Measure: Mean (Standard Deviation); unit: hours per night
Arm/Group | Amara View Minimal Contact Full Face Mask | F40 Minimal Contact Full Face Mask
Number analyzed (Participants) | 4 | 4
hours per night | 5.58 (1.35) | 4.96 (1.33)

ADVERSE EVENTS:
Time Frame: Over the one-month period that the participants were in the study (15 days per randomized mask).
Arm/Group | Amara View Minimal Contact Full Face Mask | F40 Minimal Contact Full Face Mask
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 21/35 | 25/35
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Amara View Minimal Contact Full Face Mask (N=35) | F40 Minimal Contact Full Face Mask (N=35)
Skin Irritation (Skin and subcutaneous tissue disorders) | 17 | 18
Breathing Discomfort (Respiratory, thoracic and mediastinal disorders) | 4 | 5
Aeorophagia (Gastrointestinal disorders) | 0 | 1
Knee Surgery (Musculoskeletal and connective tissue disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If PI wishes to publish study results, the Proposed Publication will be given to Philips for approval at least sixty (60) days prior to any disclosure or submission for presentation or publication. At the request of Philips, the PI agrees to (i) revise or delete any Philips' Confidential Information as requested by Philips and/or (ii) delay submission of the Proposed Publication for presentation or publication for an additional ninety (90) days to allow for filing of patient protection.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-24): https://cdn.clinicaltrials.gov/large-docs/32/NCT06535932/Prot_SAP_000.pdf